CLINICAL TRIAL: NCT07337993
Title: Efficacy of Pleural Lavage With Antifungals in the Management of Fungal Empyema Thoracis: A Prospective Cohort Study
Brief Title: Fungal Empyema Thoracis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Dr, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2025/1720/SIMS
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pyothorax; Fungal Infection Lungs; Pleural Empyema
Keywords: Fungal Pyothorax; pleural lavage; anti-fungals
MeSH Terms: conditions — Empyema, Pleural | interventions — Cerebral Decortication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pleural lavage group (Experimental): participants of this group are diagnosed as having fungal empyema on investigations of pleural fluid before any kind of surgical intervention is carried out.
  Interventions: Procedure: pleural lavage followed by surgery
- Surgical group (Active Comparator): Participants of this group are misdiagnosed as having bacterial empyema before surgery, but diagnosed as having fungal empyema intra-operatively or after surgery on post-operative culture results.
  Interventions: Procedure: Decortication
- Non-surgical group (Active Comparator): participants of this group are diagnosed as having fungal empyema and they are unfit for any kind of surgical intervention and are only managed with pleural lavage with anti-fungal drugs.
  Interventions: Other: Conservative Arm

INTERVENTIONS:
Procedure: pleural lavage followed by surgery — participants of this group are managed with pleural lavage with anti-fungals and than decortication is performed.
  Arms: pleural lavage group
Procedure: Decortication — patient underwent direct surgery for fungal empyema
  Arms: Surgical group
Other: Conservative Arm — patients are only managed with pleural lavage
  Arms: Non-surgical group

SUMMARY:
Background:

Fungal empyema thoracis is a rare but life-threatening pleural infection caused by fungal organisms such as Aspergillus and Candida species. It typically occurs in immunocompromised or debilitated patients and carries a high mortality rate. Conventional management involves systemic antifungal therapy and surgical decortication; however, many patients are unfit for surgery due to poor clinical status or multiple comorbidities. The use of local intrapleural antifungal therapy remains poorly studied.

Objective:

This study aims to evaluate the efficacy and safety of pleural lavage with voriconazole in patients with fungal empyema thoracis, both as a pre-surgical adjunct and as a palliative measure for patients who cannot undergo surgery.

Methods:

A prospective cohort study will be conducted at the Department of Thoracic Surgery, Services Hospital, Lahore. Patients diagnosed with fungal empyema confirmed by pleural fluid culture or cytology will be included. Through an indwelling chest tube, voriconazole (200 mg in 100 mL normal saline) will be instilled into the pleural cavity once daily for three consecutive days. Patients will be assessed for improvement in clinical symptoms, radiological clearance, reduction in fungal load, and the need for surgical intervention. Data will be statistically analyzed to determine treatment response and safety outcomes.

Conclusion:

Pleural lavage with voriconazole offers a promising, minimally invasive approach for managing fungal empyema thoracis. If proven effective, this method could serve as a valuable addition to current antifungal strategies, improving outcomes for critically ill patients who are not candidates for surgery.

DETAILED DESCRIPTION:
Empyema thoracis remains an important cause of morbidity and mortality worldwide. While the vast majority of pleural space infections are bacterial, fungal empyema is a distinct and increasingly recognized clinical entity that carries substantially higher mortality and a more complex therapeutic course than typical bacterial empyema. Fungal empyema most commonly occurs in patients with significant comorbidities or healthcare exposures (e.g., recent thoracic surgery, prolonged antibiotics, gastrointestinal perforation, or immunosuppression) and is frequently due to Candida or Aspergillus species. Reported crude mortality rates range between 40-70%, which are considerably higher than for bacterial empyema [1, 2].

Standard management of fungal empyema combines prompt pleural drainage with systemic antifungal therapy and, when indicated, surgical intervention (decortication or debridement) in the presence of loculation, trapped lung, or persistent sepsis [3]. However, surgical treatment is often high-risk because many patients are elderly, immunocompromised, or poor surgical candidates. Even when surgery is performed, fungal empyema is associated with increased intra- and postoperative complications and prolonged hospitalization compared with bacterial empyema [4]. These challenges underscore the need for adjunctive or alternative strategies that can enhance pleural sterilization, control sepsis, and either avert or optimize the timing of definitive surgery.

Voriconazole, a second-generation triazole antifungal, demonstrates excellent activity against Aspergillus and Candida species and has favorable pleural space penetration when administered systemically [5]. Local administration of antifungal agents directly into the pleural cavity has been described in isolated reports, with encouraging outcomes using agents such as amphotericin B and voriconazole [6-8]. Pleural lavage (intrapleural irrigation) allows high local drug concentrations at the infected pleural surface, improving fungal clearance while minimizing systemic toxicity. Case reports have demonstrated successful outcomes using intrapleural antifungal lavage as adjunct therapy or as a palliative measure in patients who could not undergo surgical decortication [7-9].

Despite these encouraging findings, there remains a paucity of prospective evidence evaluating the efficacy and safety of pleural lavage with voriconazole in fungal empyema. To address this gap, we designed a prospective cohort study to assess the outcomes of pleural lavage with voriconazole in patients with confirmed fungal empyema. The primary objectives are to evaluate (1) the effectiveness of intrapleural voriconazole lavage as an adjunct prior to surgical decortication and (2) its potential as a palliative option for patients unfit for surgery. Secondary outcomes include pleural sterilization rates, clinical improvement, conversion to surgery, length of hospital stay, and treatment-related adverse effects. This study aims to provide clinical evidence supporting the role of local antifungal therapy in optimizing the management of fungal empyema, particularly in high-risk and resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* All age patients with confirmed fungal empyema thoracis.
* Patients with adequate pleural drainage through an intercostal chest tube.
* Patients receiving systemic antifungal therapy.
* Patients either:

  1. scheduled for surgical decortication but undergoing lavage as a preoperative adjunct, or
  2. considered unfit for surgery and managed conservatively.

Exclusion Criteria:

* Bacterial empyema without fungal growth.
* Known hypersensitivity to anti-fungals.
* Severe hepatic impairment (Child-Pugh class C) contraindicating voriconazole.
* Pregnancy or lactation.
* Refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Expansion of Lung | one month post operatively
  Complete re-expansion was defined as ≥90% aeration of the ipsilateral hemithorax on postero-anterior (or AP) chest radiograph.

SECONDARY OUTCOMES:
Complications | one month post-operatively
  Post-operative complications in active surgical group and in conservative group

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, FCPS, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided